CLINICAL TRIAL: NCT02716259
Title: Impact of Basic Periodontal Therapy in the Levels of Porphyromonas Gingivalis and Aggregatibacter Actinomycetemcomitans Subgingival and Its Association With Vascular Function
Brief Title: Periodontal and Cardiovascular Diseases Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study population was insufficient to provide an adequate pool of patients. All included patients were treated and followed, but the overall desired sample size was not achieve
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Prof. Elena Figuero, Assistant Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14/120-E_BS; PI11/00542 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis; Cardiovascular Diseases
Keywords: Periodontitis; Cardiovascular diseases; Bacteremia; Scaling and root planing; Flow-mediated dilation; carotid intima-media thickness; Porphyromonas gingivalis; Aggregatibacter actinomycetemcomitans
MeSH Terms: conditions — Periodontitis; Cardiovascular Diseases; Bacteremia | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scaling and root planing (Experimental): Two sessions of scaling and root planing under local anesthesia and oral antiseptics (clorhexidine 0.12% rinse),
  Interventions: Procedure: Scaling and root planing
- Supragingival prophylaxis (Placebo Comparator): Two sessions of supragingival prophylaxis under local anesthesia and an oral rinse with no antiseptic properties.
  Interventions: Procedure: Supragingival prophylaxis

INTERVENTIONS:
Procedure: Scaling and root planing — Two sessions of scaling and root planing under local anesthesia and clorhexidine rinse twice/day, 15 days
  Other Names: Clorhexidine rinse (0.12%) (Perio-Aid, Dentaid, Spain)
  Arms: Scaling and root planing
Procedure: Supragingival prophylaxis — Two sessions of scaling and root planing under local anesthesia and sodium fluoride rinse, twice/day, 15 days
  Other Names: Sodium fluoride rinse (Fluor-Aid, Dentaid, Spain)
  Arms: Supragingival prophylaxis

SUMMARY:
The purpose of this study is to investigate whether basic periodontal therapy aim to reduce subgingival levels of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans, has an impact on the vascular function of patients suffering from established cardiovascular disease.

DETAILED DESCRIPTION:
Design: randomized clinical trial, parallel design, double blinded.

Sample: 120 patients from the Cardiology Department of Hospital Severo Ochoa (Leganés, Madrid) suffering from established cardiovascular disease and generalized moderate/severe periodontitis. Sixty patients will be randomized to test group (scaling and root planing + systemic antimicrobials), and the other 60 subjects will be included in the control group, consisting on delayed periodontal treatment (supragingival prophylaxis + placebo).

Study visits:

Visit 1: screening Visit 2: baseline data collection (medical history, clinical variables, gingival crevicular fluid (GCF) samples, vascular function) Visit 3: panoramic x-ray, blood samples, randomization and first treatment session.

Visit 4: second treatment session. Visit 5: 24 hours inflammatory biomarkers assessment. Visit 6: 7 days inflammatory biomarkers assessment. Visit 7: 1 month follow up (clinical variables) Visit 8: 3 months follow up (clinical variables, vascular function) and supportive periodontal therapy.

Visit 9: 6 months follow up (clinical variables, GCF samples, inflammatory biomarkers, vascular function) and supportive periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients with established cardiovascular disease (unstable angina or stroke in the previous 3 to 12 months, and left ventricular ejection fraction ≥50%);
* (2) diagnosis of moderate to severe generalized periodontitis (PD>5mm and marginal bone loss >30% on at least 50% of the teeth, according to Tonetti et al. 2007);
* (3) presence of at least 3 teeth per quadrant.

Exclusion Criteria:

* (1) periodontal treatment in the previous year;
* (2) antibiotic intake in the previous 3 months;
* (3) smokers of ≥10 cigarettes per day;
* (4) pregnancy or breast feeding;
* (5) diabetes mellitus types I or II, with glycosylated hemoglobin values >7;
* (6) necrotizing periodontal diseases;
* (7) HIV infection;
* (8) chronic intake of NSAID

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation of the brachial artery | Day 0 (Baseline), Day 90, Day 180
  Endothelium-dependent vasodilatation of the brachial artery assessed by means of ultrasound imaging with the use of a 7-MHz linear probe and vessel diameter measurements. Dilatation was quantified as the change in percentage form a baseline measurement and a second measurement taken after 5 minutes of flow ischemia induced with a sphygmomanometer cuff placed on the forearm.

SECONDARY OUTCOMES:
Carotid artery atherosclerosis | Day 0 (Baseline), Day 90, Day 180
  Intima-media thickness of the carotid artery assessed by means of ultrasound imaging with the use of a 7-MHz linear probe and an automated imaging software.
Periodontal pocket probing depth | Day 0 (baseline), Day 30, Day 90, Day 180
  Distance from the gingival margin to the base of the periodontal pocket, measured in 6 sites per tooth with a periodontal probe UNC-15.
Gingival recession | Day 0 (baseline), Day 30, Day 90, Day 180
  Distance from the gingival margin to the cementum-enamel junction, measured in 6 sites per tooth with a periodontal probe UNC-15.
Plaque index | Day 0 (baseline), Day 30, Day 90, Day 180
  Presence or absence of dental plaque around teeth, measured in 6 sites per tooth with a periodontal probe of the University of North Caroline (UNC)-15.
Bleeding on probing index | Day 0 (baseline), Day 30, Day 90, Day 180
  Presence or absence of bleeding 30 seconds after probing, measured in 6 sites per tooth with a periodontal probe UNC-15.
Suppuration on probing index | Day 0 (baseline), Day 30, Day 90, Day 180
  Presence or absence of gingival suppuration 30 seconds after probing, measured in 6 sites per tooth with a periodontal probe UNC-15.
Dental mobility | Day 0 (baseline), Day 30, Day 90, Day 180
  Presence of dental mobility, recorded according to Miller´s classification: 0: absence of mobility; 1: horizontal mobility <1mm; 2: horizontal mobility >1mm; 3: horizontal and vertical mobility.
Furcation lesions | Day 0 (baseline), Day 30, Day 90, Day 180
  Presence of periodontal attachment loss in the furcation area of multi-rooted teeth, recorded according to Lindhe´s classification: I: the probe penetrates less than one third of the horizontal dimension of the tooth; II: the probe penetrates more than one third of the horizontal dimension of the tooth; III: the probe penetrates through and through the tooth.
Number of present teeth | Day 0 (baseline), Day 30, Day 90, Day 180
  Number of teeth present in mouth.
Radiographic bone loss | Day 0 (baseline)
  Percentage of bone loss around teeth measured in an orthopantomography (<30%, 30-50%, >50%).
Bacteria in gingival crevicular fluid | Day 0 (baseline), Day 180
  Total counts (CFU/ml) and percentage of the flora of anaerobic bacteria present in gingival crevicular fluid. Samples will be processed by means of culture and quantitative polymerase chain reaction
Bacteria in blood samples | Day 1 (pre and post-therapy)
  Total counts (CFU/ml) and percentage of the flora of anaerobic bacteria present in blood samples before and 10 minutes after the intervention. Samples will be processed by means of culture and quantitative polymerase chain reaction
Inflammatory biomarkers in serum samples | Day 1, Day 3, Day 10, Day 180
  Levels of inflammatory biomarkers (interleukin 6, C reactive protein, e-selectin) and coagulation factors (d-dimer, prothrombin, fibrinogen, Von Willebrand factor) in serum, assessed by means of Luminex technique (Bio-Plex Pro-Assays kit).

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, Professor, Principal Investigator — Faculty of Dentistry, Complutense University of Madrid; David Herrera, Professor, Principal Investigator — Faculty of Dentistry, Complutense University of Madrid; Elena Figuero, Professor, Study Director — Faculty of Dentistry, Complutense University of Madrid; María Molina, Doctor, Study Chair — Servicio de Cardiología, Hospital Universitario Severo Ochoa
Locations (2):
- Spain (2):
  - Severo Ochoa Hospital, Leganés, Madrid
  - Faculty of dentistry, Complutense University Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Derived] Molina A, Ambrosio N, Molina M, Montero E, Virto L, Herrera D, Figuero E, Sanz M. Effect of periodontal therapy on endothelial function and serum biomarkers in patients with periodontitis and established cardiovascular disease: a pilot study. Front Oral Health. 2025 Feb 10;6:1488941. doi: 10.3389/froh.2025.1488941. eCollection 2025. PMID 39996093